CLINICAL TRIAL: NCT02810483
Title: Randomized, Placebo Controlled Double-blind Study of the Efficacy of Topiramate on the Symptoms of Irritability - Impulsivity, Overeating and Self-harm in a Population of Patients Suffering From Prader Willi Syndrome Over 8 Weeks
Brief Title: Study of the Efficacy of Topiramate in Patients With Prader Willi Syndrome Over 8 Weeks
Acronym: TOPRADER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AOM10088
Record Dates: First submitted 2016-05-17; First posted 2016-06-23 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2016-04

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi; SPW; impulsivity; eating disorders; topiramate
MeSH Terms: conditions — Prader-Willi Syndrome; Impulsive Behavior; Feeding and Eating Disorders | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Topiramate (Experimental): Topiramate Arrow 50 mg hard capsules
  Interventions: Drug: Topiramate
- Arm 2: Placebo Comparator (Placebo Comparator): 50 mg hard capsules with the same shape, color and taste than the active product
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Topiramate — Increase phase. The starting dose is 50 mg / day with gradual increase in dose to 50 mg / week until the end of the 3rd week.
  Dose of study:
  200mg for 5 weeks.
  Decrease phase:
  The 9th week, 100mg for 4 days then 50mg for 3 days.
  Other Names: Topiramate Arrow generic
  Arms: Arm 1: Topiramate
Drug: Placebo Comparator — ncrease phase. The starting dose is 50 mg / day with gradual increase in dose to 50 mg / week until the end of the 3rd week.
  Dose of study:
  200mg for 5 weeks.
  Decrease phase:
  The 9th week, 100mg for 4 days then 50mg for 3 days.
  Arms: Arm 2: Placebo Comparator

SUMMARY:
There is no specific treatment for core symptoms of PWS. Regarding behavioral and psychiatric symptoms (hyperphagia, imulsivity and self-mutilations), one of the only drug options consists in antipsychotics, that are not efficient and might be responsible for a worsening of the weight gain (major issue in PWS). An alternative therapeutic approach for behavioral disturbances has been suggested by some authors with topiramate (Epitomax®), an antiepileptic drug that can be used as a mood stabilizer and anti-impulsive. In addition, topiramate is used as a treatment for eating disorders because it induces loss of weight and appetite. This last effect might be useful in the case of SPW.

Except for some clinical case reports, the investigators only found one open study for topiramate in SPW 8 patientssuggesting promising effects. There si however no placebo controlled study..

Objective:

To evaluate the efficacy of topiramate (200 mg / d) on Eating disorders (E), self Mutilations (M), irritability and Impulsivity (I), metabolic status, and tolerance among of PWS patients.

Methodology:

This is a multicenter (out-patients in Toulouse, Reims, Nantes and Paris and in-patients in Hendaye) 8 weeks double-blind placebo controlled study .

Subjects (n = 125 for 112 analyzable) all having PWS, aged 12 years-old and more should have any of the following symptoms: E, M and U (see above). All subjects will be randomly allocated into two groups one taking a placebo, the other taking topiramate (50mg / day initially, increasing up to 50mg per week 200mg / day).

The population of analyzable patients in and out patient will be of equal size (n = 56). The inclusion period is two years..

Are excluded subjects with antipsychotic or mood stabilizer medication or topiramate.

The primary endpoint will be the rate of responders, with response defined by obtaining a score of 1 or 2 on the CGI improvement after 8 weeks of treatment

Other assessments, secondary endpoints :

* Clinic: Weight / Size / Self-injury behavior (french Echelle des Conduites Auto et Hétéro Aggressives, ECAHA))
* Psychometric: C-SHARP and A-SHARP / Conners (Impulsivity) / Dickens (Eating behavior for PWS)
* Organic: NFS, serum electrolytes, creatinine, ammonia plasma, serum bicarbonate, AST / ALT / GGT, ghrelin, fasting glucose, lipid profile and insulin, leptin, TG and HbA1c.
* Side effects of topiramate: SAPS / SANS and BPRS (hallucinations), anxiety scales and laboratory tests.

DETAILED DESCRIPTION:
Scientific background and justification of the study :

Patients with a rare disease are often challenging to treat when considering psychotropic treatment for behavioral or psychiatric manifestations. There is an important lack of clear data or treatment guidelines for treating behavioral disturbance in patients with intellectual disabilities. Prader Willi syndrome (PWS) is a paradigmatic example of such a disease. It is a rare disease with an estimated prevalence of 1:25,000 at birth. PWS is a genetic disease located on chromosome 15 (15 q11-q13). Imprinting silence the normal genes on 15 q11-Q13, rendering them non-functional, with the paternal non-imprinted genes being deleted. The imprinting effect in this region explains why approximately 60 to 70% of patients with PWS have a paternal deletion of 15q11-q13 (2). An additional 25 to 35 % of patients have two copies of maternal chromosome 15 (uniparental disomy). Rarely, PWS may be associated with translocation, mutation, or other anomalies. Angelman Syndrome, which has primarily been associated with autism spectrum disorders, involves the same genetic region and is commonly associated to mutations of the maternal allele of the UB3a gene or rare deletions. .

PWS patients present in a neonatal hypotonic state with deficit of sucking and eating refusal which progresses to with hyperphagia and obsession with food in infancy or adolescence. In addition, patients have distinct facial features, such as a narrow forehead, almond-shaped eyes, and a triangular mouth, as well as a short stature, related to growth hormone deficiency and small hands and feet. Puberty is often delayed or incomplete, and most affected individuals are unable to have children. This eating disorder is more similar to an addictive disorder to food than a traditional eating disorder. PWS leads to severe obesity, which is a major issue associated with quality of life and medical prognosis.

Psychiatric and cognitive symptoms in patients with PWS are severe and have an important impact on social and interpersonal life. Patients with PWS often have mild to moderate intellectual disability (ID), with learning impairments and poor academic achievement. They have particular difficulties in mathematics, calculation, and abstraction, which may be related to under-diagnosed neuro-visual impairments. There is a large individual heterogeneity of language impairments, primarily in morphosyntaxic abilities. Behavioral impairments predominately include temper outbursts, impulsivity, emotional liability and aggressive behavior , as well as self-injury behavior, such as compulsively picking the skin and mucosa (rectal picking), which may lead to a severe wound and severe infections. Patients with disomy as a group have more severe overall symptoms than patients with a deletion.

Regarding the relationship between PWS and schizophrenia spectrum disorders (SSDs), 5 studies have utilized standardized psychometric tools to assess psychiatric diagnoses. SSDs are primarily, but not exclusively, associated with disomy, and the clinical diagnosis may be complicated. Considering that disomy represents only 20%, at most, of patients, SSDs affect less than 20% of patients with PWS, most likely approximately 17% or 15%. There are few studies in the field of behavioral treatment in PWS they suggests that risperidone for psychotic symptoms associated with disomy, and N-acetylcysteine for skin picking might be efficient. Moreover and despite many study limitations, the investigators identified promising treatment effects with topiramate for self-injury and impulsive/aggressive behaviors. To date there is only one study (open trial) for topiramate in PWS.

Our aim is to assess efficacy and tolerance of topiramate in behavioral disturbance in patients with PWS.

Main objective :

Assess the efficacy and tolerance of topiramate at 200 mg / day on hyperphagia (H), seflf-injury (SI) and Irritability-Impuslivity Behavior in patients with Prader Willi Syndrome during an 8 weeks follow-up.

Secondary objective Assess the tolerance and side effect ot topiramate 200mg/day in this specific population.

Methodology :

The investigators will run a multicentric double blind placebo controlled randomized trial with outpatients in Paris and Toulouse and inpatients in Hendaye. Inclusion period is 3 years in order to obtain a total number of participants of 125 randomly assigned in two groups (drug vs placebo).

Local Ethic Committee did approve this research. Patients and/or their parents / caregiver give informed consent.

Main outcome measure will be Clinical Global Impression thereshold will be to obtain at least 1 at CGI Improvement scoring at endpoint after 8 weeks follow-up.

Secondary outcome (psychometric scales and biological measures):

* Weight, Self-Injury Behavior, C-SHARP and A-SHARP (suicide ideation scale, according to age), CONNERS Impulsivity, Dickens (Hyperphagia)
* Sides effects assessment; PANNS (for hallucinations), Eysenck Anxiety
* And biological assessment including lipid, hepatic enzyme, insulin, serum bicarbonate, leptin, amoniemia, ghreline and HbA1c.

Instruments and assessments. Psychometric scales: Impulsivity and aggressive behavior will be evalauated with irritability sub-score of Aberrant Behaviour Checklist The Children's Scale of Hostility and Aggression: Reactive/Proactive (C-SHARP) for adolescents until 16 years-old and The Adult Scale of Hostility and Aggression: Reactive/Proactive (A-SHARP) for adults. The Dickens questionnaire, especially oriented for PWS patients, will be used for eating behavior. Self injury behavior will be assessed with Scale of Self-Aggressive Behavior (ECAA Yale-Paris), especially in the sub -scale regarding severity, duration and frequency of such behavior. The Clinical Global Impression, will be used at base line, 2, 4, 6 and 8 weeks (endpoint).

Scale for the Assesment of Positive Symptoms, SAPS, and Brief Psychiatric Rating Scale, BPRS, Hamilton Anxiety Sclale, HAS et Columbia Classification Algorithm of Suicide Assessment (C-CASA).

Somatic assessment: Blood sample with routine elements associated with complete blood count, creatinin, amoniemia serum bicarbonate, ASAT/ALAT/γGT, glycemia lipid profil and insulin, ghrelin, leptin, TG and HbA1c. Weight and size in order to calculate the Body Mass Index. Centralized blood level of drug concentration at baseline (no treatment), week 4 and week 8.

Design and timeline :

Selection will be made on inclusion/exclusion criteria including blood sample. Inclusion and randomization is at baseline and all assessments will be made.

Visits are scheduled at week 2, 4, 6 and 8 (endpoint and end of patient participation). All scales are used for all visit and biological sample are made at selection, inclusion, week 4 and week 8.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with Prader Willi syndrome confirmed by genetic diagnosis.
2. Patient has at least one of the following symptoms:

   * Presence of self-harm
   * Impulsive and / or aggressive
   * Trouble eating and / or obesity
3. Age between 12 and 45 years inclusive
4. Weight higher than 50 kg
5. Signature of consent by the patient or the holders of parental authority (or legal guardian)

Non inclusion criteria:

1. Meeting the criteria according to DSM IV Schizophrenia
2. Presence of hallucination (SAPS scales and scale of hallucination)
3. Already has an effective dose of topiramate for a sufficient time and without efficiency
4. Psychotropic introduced for less than three months or dose change for less than three months.
5. Psychotropic stopped for less than a month, or three months in the case of fluoxetine.
6. Inability to find an informative adult in the subject's behavior.
7. Known hypersensitivity to one of topiramate constituents or its placebo
8. Known hypersensitivity to sulfonamides
9. Epilepsy associated or taking other anticonvulsant or mood stabilizer.
10. Medication with St. John's wort
11. No affiliation to a social security
12. Patient known to be non-compliant
13. Subject to suicide risk
14. Severe depression
15. Previous history of nephrolithiasis or glaucoma
16. Poorly controlled diabetes (A1C greater than 10%) treated with metformin or Gibenclamide.
17. Patients with rare hereditary problems of fructose intolerance, glucose malabsorption or galactose or sucrose-isomaltase insufficiency (because of the presence of sucrose)
18. Pregnant or breastfeeding
19. Lack of effective contraception among patients of childbearing potential

Exclusion criteria before randomization:

* Renal failure (serum creatinine greater than 1.5 X normal)
* Hepatic impairment (ALT greater than 2X normal) (
* Anemia (HB <12 g / dl female <13g / dl man.)
* Hyper ammonemia (upper normal laboratory)
* Responding to the Schizophrenia criteria according to DSM IV
* Presence of hallucination (SAPS scales and scale of hallucination)
* Decreased serum bicarbonate levels (below the laboratory standards)

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2012-12; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Improvement | at 8 weeks (endpoint)
  Endpoint CGI score at 1 or 2 will make consider the patient as a responder. A 7 items scale will be used

SECONDARY OUTCOMES:
Weight and size | at 8 weeks (endpoint)
  Weight and size (BMI in kg/m2)
Self-Injury Behavior Scale ECAHA, | at 8 weeks (endpoint)
  Comparison between baseline score and endpoint score
Self-Injury Behavior, CONNERS Impulsivity | at 8 weeks (endpoint)
  CONNERS Impulsivity comparison between baseline score and endpoint score
Self-Injury Behavior,Dickens | at 8 weeks (endpoint)
  Dickens comparison between baseline score and endpoint score
C-SHARP (Chid and Adolescent), appearance of positive suicide item response | at 8 weeks (endpoint)
A-SHARP (Adult), appearance of positive suicide item response | at 8 weeks (endpoint)
  A-SHARP (Adult), appearance of positive suicide item response
Safety Assessment | at 8 weeks (endpoint)
  The proportion of patients stopped the treatment, of patients with adverse events and prematurely discontinued treatment due to an adverse event will be estimated.
Biological assessment | at 8 weeks (endpoint)
  The number of patients with abnormal values and / or modified from the baseline values will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BONNOT, PhD, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital La Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No